CLINICAL TRIAL: NCT04804839
Title: Comparison of the Effectiveness of Different Conservative Treatment Protocols in Individuals With Symptom of Postprostatectomy Urinary Incontinence : a Randomized Controlled Trial
Brief Title: Comparison of the Effectiveness of Different Conservative Treatment Protocols in Postprostatectomy Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-20081
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence; Prostate Cancer; Urinary Incontinence,Stress; Urinary Incontinence Due to Urethral Sphincter Incompetence
Keywords: Knack maneuver; Pelvic floor muscle training; Lifestyle interventions; Kegel exercises; Prostate cancer; Men's health; Pelvic floor exercises
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms; Urinary Incontinence, Stress | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First research arm (Combined group) (Experimental): Combined group with 8 weeks of pelvic floor muscle training, knack maneuver and lifestyle recommendations.
  Interventions: Other: First research arm
- Second research arm [PFMT (including knack maneuver) group] (Experimental): Only 8-week PFMT (including knack maneuver)
  Interventions: Other: Second research arm
- Third research arm (PFMT alone group) (Active Comparator): It is the control group and patients in this group were given alone8-week PFMT (without knack maneuver).
  Interventions: Other: Third research arm

INTERVENTIONS:
Other: First research arm — Patients in this group were given 8-week PFMT (including knack maneuver) and lifestyle recommendations for the treatment of urinary incontinence symptoms.
  Other Names: Combined group
  Arms: First research arm (Combined group)
Other: Second research arm — Patients in this group were given only 8-week PFMT (including knack maneuver) for the treatment of urinary incontinence symptoms.
  Other Names: PFMT (including knack maneuver) group
  Arms: Second research arm [PFMT (including knack maneuver) group]
Other: Third research arm — It is the control group and patients in this group were given alone8-week PFMT (without knack maneuver).
  Other Names: PFMT alone group
  Arms: Third research arm (PFMT alone group)

SUMMARY:
The main purpose of this study is to reveal the effectiveness of the Knack maneuver and lifestyle recommendations program to be given in addition to the pelvic floor muscle training (PFMT) program, which has been proven to be effective in individuals with urinary incontinence symptoms after prostatectomy. This study is a prospective, controlled, randomized clinical trial. The study includes an 8-week pelvic floor muscle training, Knack maneuver and lifestyle recommendations.

In summary, it is stated in the literature that PFMT and lifestyle recommendations are beneficial in the treatment of urinary incontinence (UI). However, although there is evidence of the effectiveness of the Knack maneuver in stress UI in women, there is no evidence of the Knack maneuver in urinary incontinence after prostatectomy. On the other hand, the literature on the effect of lifestyle recommendations after prostatectomy is very limited.

Therefore, the aim of this study is to reveal the effectiveness of the Knack maneuver and lifestyle recommendations program, which will be given in addition to the PFMT program, which has been demonstrated in individuals with UI complaints after radical prostatectomy, in a randomized controlled design.

DETAILED DESCRIPTION:
The main purpose of this study is to reveal the effectiveness of the Knack maneuver and lifestyle recommendations program to be given in addition to the pelvic floor muscle training (PFMT) program, which has been proven to be effective in individuals with urinary incontinence symptoms after prostatectomy. This study is a prospective, controlled, randomized clinical trial. The study includes an 8-week pelvic floor muscle training, Knack maneuver and lifestyle recommendations.

It was planned to enroll 72 individuals with urinary incontinence problems after radical prostatectomy in this randomized controlled clinical study. A physical therapist is responsible for all assessments.

Participants were included in one of three treatment groups (G1: Pelvic floor muscle training + Knack maneuver + lifestyle recommendations; G2: Pelvic floor muscle training + Knack maneuver G3: Pelvic floor muscle training).

In summary, it is stated in the literature that PFMT and lifestyle recommendations are beneficial in the treatment of urinary incontinence (UI). However, although there is evidence of the effectiveness of the Knack maneuver in stress UI in women, there is no evidence of the Knack maneuver in urinary incontinence after prostatectomy. On the other hand, the literature on the effect of lifestyle recommendations after prostatectomy is very limited.

Therefore, the aim of this study is to reveal the effectiveness of the Knack maneuver and lifestyle recommendations program, which will be given in addition to the PFMT program, which has been demonstrated in individuals with UI complaints after radical prostatectomy, in a randomized controlled design.

With this study, the effectiveness of different programs to be applied to individuals suffering from urinary incontinence after prostatectomy will be determined and compared. It will increase the level of evidence for the treatment of urinary incontinence, a common complaint after prostate cancer surgery. In this direction, it will also contribute to the development of public health.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18 years of age (with a Mini Mental Test score ≥ 24 for individuals over the ages of 65), who had a complaint of UI after prostatectomy, who did not have any cooperation problems in the evaluations or practices in the study, were included.

Exclusion Criteria:

* Acute disease state (e.g. urinary tract infection, upper respiratory tract infection, interstitial cystitis, bladder or gastrointestinal bleeding), acute surgical condition (occurring within the first 3 weeks after prostatectomy), neurological disease, or participants with neurogenic bladder, participants with complaints of pure urgency urinary incontinence, presence of preoperative incontinence, who have undergone bladder or other prostate surgeries prior to prostatectomy, who did not give consent to the study and who do not have an informed consent form will not be included.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be conducted in patients suffering from urinary incontinence after prostatectomy.
Enrollment: 72 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Modular Questionnaire - Urinary Incontinence short form (ICIQ-UIsf (short form)) | In the first evaluation(baseline), during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Symptom severity and impact of incontinence on life

SECONDARY OUTCOMES:
Patient Global Impression of Severity question | In the first evaluation(baseline), during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Individual's perception of symptom severity
1 hour pad test | In the first evaluation(baseline), during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Incontinence severity Pad Test assesses urine loss and leakage volume of the participant
King's Health Questionnaire | In the first evaluation(baseline), during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Impact of incontinence on quality of life
Patient Global Impression of Improvement question | Post-treatment evaluation (at the end of the eighth week)
  Individual's perception of improvement

OTHER OUTCOMES:
International Physical Activity Questionnaire and Likert-type scales. | During study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Compliance with lifestyle change recommendations
Likert-type scales | during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Compliance with smoking, alcohol, tea, caffeine, carbonated beverage, water consumption, bowel order management, exercise and physical activity recommendations will be evaluated separately.
Exercise diary | during study (at the end of the fourth week), post-treatment evaluation (at the end of the eighth week)
  Adherence to the home exercise program will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Kaya, Assoc Prof, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerlegiz ENA, Akbayrak T, Gursen C, Yazici MS, Bolat NM, Akdogan B, Nakip G, Ozgul S. Lifestyle recommendations and pelvic floor muscle training with Knack maneuver for post-prostatectomy urinary incontinence: a randomized controlled trial. Support Care Cancer. 2025 Jan 31;33(2):132. doi: 10.1007/s00520-025-09197-z. PMID 39888446